CLINICAL TRIAL: NCT05563649
Title: Confirming the Effectiveness and Efficiency of Online Guided Self-Help Family-Based Treatment for Adolescent Anorexia Nervosa
Brief Title: Confirming the Effectiveness of Online Guided Self-Help Family-Based Treatment for Adolescent Anorexia Nervosa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James Dale Lock, Professor of Child Psychiatry and Pediatrics in the Department of Psychiatry and Behavioral Sciences and Director of the Eating Disorder Program for Children and Adolescents, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 67295; R01MH130388 (NIH)
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online Guided Self-Help-Family-based Treatment (GSH-FBT) (Experimental): GSH-FBT consists of 10 20-minute parent-only sessions over 9 months. The guidance portion is manualized and will be delivered by a clinician familiar with both the online modules and FBT, who acts as a "coach." Sessions follow an online curriculum containing a total of 65 short videos. Each lecture series is comprised of a written introduction orienting the viewer to the videos, 5-9 short videos (< 7 minutes each), and assigned reading from the parent education manual, Help Your Teenager Beat an Eating Disorder. In line with GSH approaches, coaches direct parents to watch or re-watch specific videos contained in the online platform related to their questions.
  Interventions: Behavioral: Online Guided Self-Help-Family-based Treatment
- FBT via Videoconferencing (FBT-V) (Active Comparator): 15 60-minute sessions of 3-phase manualized FBT modified for videoconferencing will be delivered to participants randomized to this treatment by therapists trained in FBT. The first phase encourages parental management of weight restoration (approximately 8 weekly sessions); the second phase promotes a developmentally appropriate transition back to adolescent management of weight restoration and maintenance under parental supervision (approximately 4 bi-weekly sessions), and the third phase focuses on adolescent development (approximately 3 monthly sessions). Each session consists of 10 minutes with the adolescent individually to discuss progress and the adolescent's perspective on treatment, followed by 50 minutes with the entire family.
  Interventions: Behavioral: FBT via Videoconferencing

INTERVENTIONS:
Behavioral: Online Guided Self-Help-Family-based Treatment — GSH-FBT consists of 10 20-minute sessions for parents only over 9 months. Sessions follow an online curriculum of 65 short videos: 62 with an expert clinician instructing parents on the principles of FBT, and 3 reflections from an adolescent who recovered from AN and completed FBT. Each lecture series contains an introduction orienting the viewer to the videos, 5-9 short videos (< 7 minutes each), and assigned reading from the parent education manual Help Your Teenager Beat an Eating Disorder. Three lectures include additional resources for parents (e.g., Academy of Eating Disorder (AED) Medical Management Guidelines). Homework assignments are included with some lectures (e.g., strategies to help the child eat during meals, practice making calorically dense meals). In line with GSH approaches, coach-therapists direct parents, to watch or re-watch specific video content contained in the online learning material related to their questions rather than direct behavioral change.
  Other Names: GSH-FBT
  Arms: Online Guided Self-Help-Family-based Treatment (GSH-FBT)
Behavioral: FBT via Videoconferencing — 15 60-minute sessions of 3-phase manualized FBT modified for videoconferencing will be delivered to participants randomized to this treatment by therapists trained in FBT. The first phase encourages parental management of weight restoration (approximately 8 weekly sessions); the second phase promotes a developmentally appropriate transition back to adolescent management of weight restoration and maintenance under parental supervision (approximately 4 bi-weekly sessions), and the third phase focuses on adolescent development (approximately 3 monthly sessions). Each session consists of 10 minutes with the adolescent individually to discuss progress and the adolescent's perspective on treatment, followed by 50 minutes with the entire family.
  Other Names: FBT-V
  Arms: FBT via Videoconferencing (FBT-V)

SUMMARY:
With an incidence rate of about 1%, Anorexia Nervosa (AN) is a serious mental disorder associated with high mortality, morbidity, and cost. AN in youth is more responsive to early treatment but becomes highly resistant once it has taken an enduring course. The first-line treatment for adolescents with AN is Family Based Treatment (FBT). While FBT can be delivered using videoconferencing (FBT-V), therapists' limited availability hampers scalability. Guided self-help (GSH) versions of efficacious treatments have been used to scale and increase access to care. The main aim of this proposed comparative effectiveness study is to confirm that clinical improvements in GSH-FBT are achieved with greater efficiency than FBT-V in generalizable clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are 12-18 years of age
2. Participants live with a family (some families may contain only one parent)
3. Family members fluently speak and read English and have access to a computer with internet
4. Participants meet DSM-5 criteria for AN (both subtypes)
5. EBW above 75%
6. Participants are medically stable for outpatient treatment according to the recommended thresholds of the American Academy of Pediatrics and the Society of Adolescent Medicine
7. Participants are not engaged in another individual or family-based psychotherapy trial during the duration of treatment sessions in the study.
8. Medications for comorbid psychiatric disorders are OK; randomization will balance groups through tracking.

Exclusion Criteria:

Current psychotic illness or intellectual disability or other mental illnesses that would prohibit the use of psychotherapy; current dependence on drugs or alcohol; physical conditions (e.g. diabetes mellitus, pregnancy) known to influence eating or weight; previous FBT; and inability of the participant and/or family to speak and understand English.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Ratio of therapist hours to %EBW change | Assessed from baseline through end of treatment (EOT)
  The investigators will compare GSH-FBT and FBT-V groups at EOT in terms of the change in %EBW from baseline divided by total therapist time utilized. Estimated Body Weight (EBW) percentages used will be calculated using Center for Disease Control metrics in children and adolescents. Total therapist time utilized will be collected based on video records of actual sessions spent with participants.

SECONDARY OUTCOMES:
Eating Disorder Examination (EDE) | Baseline (before beginning treatment); 3 months within treatment; 9 months (EOT); and at 6- and 12-month follow-up
  The EDE is a standardized investigator-based interview that measures the severity of the characteristic psychopathology of eating disorders. The psychometric properties of the EDE are sound and validated in diverse samples. It takes about 1 hour to complete.
Beck Depression Inventory (BDI) | These assessments will be collected bi-weekly (sessions 2, 4, 6, 8) and at all major assessment points (BL, 3 months within treatment, EOT, 6 and 12-month follow-up)
  The BDI is a measure with sound psychometric properties and was validated on a diverse sample. It has been used in numerous studies of adolescent depression. This measure also includes questions about suicidal ideation and intent and will be used to assess suicide during the study. These assessments will be collected bi-weekly (sessions 2, 4, 6, 8) and at all major assessment points. It takes about 10 minutes to complete.
Beck Anxiety Inventory (BAI) | Baseline, sessions 2, 4, 6, 8, and EOT
  The BAI is a 21-item questionnaire about anxiety that has sound psychometric properties and was validated on a diverse sample. Assessments will be collected at baseline, sessions 2, 4, 6, 8, and EOT.

CONTACTS AND LOCATIONS:
Locations (2):
- Stanford University, Stanford, California, United States
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No